CLINICAL TRIAL: NCT06517407
Title: Para Rectus Versus Trans Rectus Stoma Placement for Prevention of Stoma Related Complications
Brief Title: Para Versus Trans Rectus Stoma Placement for Prevention of Stoma Related Complications
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Sayed Mohamed Sayed, General surgery department at assiut university Hospitals, Assiut University
Other Study IDs: Stoma placement
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Stoma Malfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fecal divertion is a surgical procedure by which stoma is constructed through exteriorization of small intestine or large intestine(loop or end stoma).There are many indications for enterostomies such as malignancy, bleeding per rectum, MVO, Volvulus, iatrogenic colon injury, adhesive bands....... etc.

Many factors concerning the operative technique are considered to influence the incidence of stoma related complications such as stoma prolapse, retraction, stenosis, para stomal herniation, para stomal soiling ,oedema and ileus. Site of stoma creation in relation to rectus abdominis muscle is believed to be one of them.

DETAILED DESCRIPTION:
Fecal divertion is a surgical procedure by which stoma is constructed through exteriorization of small intestine or large intestine(loop or end stoma).There are many indications for enterostomies such as malignancy, bleeding per rectum, MVO, Volvulus, iatrogenic colon injury, adhesive bands.

Many factors concerning the operative technique are considered to influence the incidence of stoma related complications such as stoma prolapse, retraction, stenosis, para stomal herniation, para stomal soiling ,oedema and ileus. Site of stoma creation in relation to rectus abdominis muscle is believed to be one of them.

ELIGIBILITY:
Inclusion Criteria:

* All patient who recieve abdominal enterostomies either elective or emergencies in surgery department of assuit university hospital

Exclusion Criteria:

1. Patient underwent repair of previous abdominal surgery
2. Patient known to have incisional or ventral abdominal hernia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lateral para rectal or trans rectal stoma exteriorization.
  * Stoma site was incised about 3-5 cm from lateral edge of rectus abdominal muscle at para rectus position, or
  * at he lateral edge of the rectus abdominal muscle in trans rectal position
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
para stomal herniation | 6 months
  * Stoma site was incised about 3-5cm from lateral edge of rectus abdominis muscle at para rectus position, or
  * at he lateral edge of the rectus abdominis muscle in trans rectal position.

SECONDARY OUTCOMES:
a_wound infection b_post operative ilieus c_oedema of the stoma d_soiling around the stoma e:prolapse f: stenosis g:retraction | 6 months
  Stoma related other complication

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hardt J, Meerpohl JJ, Metzendorf MI, Kienle P, Post S, Herrle F. Lateral pararectal versus transrectal stoma placement for prevention of parastomal herniation. Cochrane Database Syst Rev. 2019 Apr 24;4(4):CD009487. doi: 10.1002/14651858.CD009487.pub3. PMID 31016723